CLINICAL TRIAL: NCT00555438
Title: Prospective, Multicentre, Open-label Study Evaluating 1.5 mg/Day of Fondaparinux,in Venous Thromboembolic Events Prevention in Patients With Renal Impairment and Undergoing a Major Orthopaedic Surgery. PROPICE Study
Brief Title: Prospective, Multicentre, Open-label Study Evaluating 1.5 mg/Day of Fondaparinux.
Acronym: PROPICE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Pr Patrick MISMETTI, Centre Hospitalier Universitaire de Saint Etienne
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0701017; 2007-001048-32 (EudraCT Number)
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Results first posted 2010-11-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-07

CONDITIONS: Major Orthopaedic Surgery and Renal Impairment
Keywords: major orthopaedic surgery; venous thromboembolic events prevention; renal impairment; Arixtra; anti-Xa activity
MeSH Terms: conditions — Renal Insufficiency | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): patients with renal impairment who received Fondaparinux 1.5 mg/l after major orthopaedic surgery
  Interventions: Drug: fondaparinux 1.5 mg/day

INTERVENTIONS:
Drug: fondaparinux 1.5 mg/day — Subcutaneous injection of fondaparinux 1.5 mg/l after major orthopaedic surgery

SUMMARY:
Fondaparinux is an antithrombotic agent having already received a regulatory approval by the European Authorities in venous thromboembolic event prevention after major orthopaedic surgery, as total hip replacement (THR), total knee replacement (TKR), hip fracture (HF). The bleeding risk associated with this prescription is highly related to renal function evaluated by creatinin clearance (CrCl). In order to reduce the bleeding risk, it has been proposed to prescribe fondaparinux 1.5 mg/day in patients with a CrCl between 20 and 50ml/mn instead of 2.5mg/day (European MMA). In the meantime, this approval is essentially based on simulated pharmakinetic data without any support of clinical data.

prospective, multicentre, open-label study evaluating the safety profile of fondaparinux 1.5 mg/day, subcutaneously administered, in patients with a renal impairment defined by a CrCl between 20 and 30 ml/min and undergoing a major orthopaedic surgery.

DETAILED DESCRIPTION:
Fondaparinux 1.5mg/day subcutaneously administered during post-surgery 1 to 10 days with the 1st treatment administration performed 6 to 8 hours after the end of surgery.

Screening visit : > 7 days before inclusion visit if THR and TKR Inclusion visit : day of surgery Visits with blood drawing: 3 visits scheduled during 1 to 10 days of treatment period Study end of treatment visit: D1 to D10 Study end visit: 1 month ± 15 days

ELIGIBILITY:
Inclusion Criteria:

* • age > 18 years old,

  * undergoing a major orthopaedic surgery (THR, TKR, HF) whatever procedure techniques are used, 1st indication or 2nd indication,
  * requiring an antithrombotic prophylaxis,
  * presenting a renal impairment defined by a creatinin clearance (CrCl) between 20 and 50 ml/min calculated by Cockcroft and Gault's formula,
  * having signed the inform consent form.

Exclusion Criteria:

* contra-indications to fondaparinux,
* history of heparin inducted thrombopenia (HIT),
* platelets < 100 g/l.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MISMETTI Patrick, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (29):
- France (29):
  - GARANGER Thierry, Agen
  - CHARRET Françoise, Annonay
  - BONNEMAISON Julie, Bayonne
  - BELLOUCIF Sadek, Bobigny
  - SZTARCK François, Bordeaux
  - PEGOIX Michel, Caen
  - AUSSET Sylvain, Clamart
  - SCHOEFFLER Pierre, Clermont-Ferrand
  - LETOURNEAU Bernard, Dijon
  - TISSIER Dominique, La Roche-sur-Yon
  - LEMANISSIER Denis, Le Mans
  - CHAMBON Françoise, Lyon
  - BEGOU Gérard, Lyon
  - CAPDEVILLA Xavier, Montpellier
  - PERON Alain, Nantes
  - GAERTNER Elisabeth, Nice
  - CHEVALEREAUD Erick, Niort
  - RIPART Jacques, Nîmes
  - LANGERON Olivier, Paris
  - RABUEL Christophe, Paris
  - MAZUIRE Elisabeth, Paris
  - THERY Philippe, Poitiers
  - BARRE Jeanne, Reims
  - LIGNOT Sophie, Rouen
  - MARTIN, Saint-Etienne
  - BAYLOT Denis, Saint-Etienne
  - DUVERGER Daniel, Saint-Saulve
  - FUZIER Régis, Toulouse
  - COUVRET Claude, Tours

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients have been included between june 2007 and june 2008 in public and private French hospitals
Pre-assignment Details: Nine patients received no study drug due to immediate postoperative death (n=1), consent withdrawal (n=2), use of another thromboprophylactic agent (n=2), surgery change or cancellation (n=2), and CrCl >50 mL/min just before surgery (n=2)
Groups:
- Fondaparinux 1.5 mg/l: patients with renal impairment who received Fondaparinux 1.5 mg/l after major orthopaedic surgery
Period: 10 Days Post-operative
Arm/Group | Fondaparinux 1.5 mg/l
Started | 442
Completed | 438 (438 patients attended the day 10 visit (four patients died during hospitalization))
Not Completed | 4
Not completed — Death | 4
Period: Between 10 Days and 30 Days Postoperativ
Arm/Group | Fondaparinux 1.5 mg/l
Started | 438
Completed | 433
Not Completed | 5
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Arm/Group | Fondaparinux 1.5 mg/l
Number analyzed (Participants) | 442
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 437
Age Continuous [Mean (Standard Deviation); unit: years] | 81.4 (6.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 353
  Male | 89
Region of Enrollment [Number; unit: participants]
  France | 442

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Major Bleedings Between Day 1 and Day 10.
Description: evaluate between Day 1 and Day 10, the number of patients under study treatment who has affected by major bleedings defined as fatal, involved a critical organ, treatment cessation, occurred at the surgical site and necessitated any medical intervention, or if it was overt and necessitated transfusion of >2 units of packed red blood cells or was associated with a fall in hemoglobin >20 g/L.
Time Frame: 10 day
Measure: Number; unit: participants
Arm/Group | Fondaparinux 1.5 mg/l
Number analyzed (Participants) | 442
participants | 20

2. Secondary Outcome: Number of Patients With Major Bleedings at 1 Month ± 5 Days.
Description: evaluate the number of patients affected by major bleedings defined as fatal, involved a critical organ, treatment cessation, occurred at the surgical site and necessitated any medical intervention, or if it was overt and necessitated transfusion of >2 units of packed red blood cells or was associated with a fall in hemoglobin >20 g/L at 1 month ± 5 days.
Time Frame: 45 day
Measure: Number; unit: participants
Arm/Group | Fondaparinux 1.5 mg/l
Number analyzed (Participants) | 442
participants | 23

3. Secondary Outcome: Number of Patients With Symptomatic Deep Vein Thrombosis and Pumonary Embolism Between Day 1 and Day 10
Description: Evaluate the number of patients affected by symptomatic Deep Vein Thrombosis (any symptomatic distal and/or proximal deep-vein thrombosis) and Pumonary Embolism (symptomatic pulmonary embolism confirmed by objective tests) between Day 1 and Day 10.
Time Frame: 10 days
Measure: Number; unit: participants
Arm/Group | Fondaparinux 1.5 mg/l
Number analyzed (Participants) | 442
participants | 2

4. Secondary Outcome: Number of Patients With Symptomatic Deep Vein Thrombosis and Pumonary Embolism at 1 Month ± 5 Days
Description: Evaluate the number of patients affected by symptomatic Deep Vein Thrombosis (any symptomatic distal and/or proximal deep-vein thrombosis) and Pumonary Embolism (symptomatic pulmonary embolism confirmed by objective tests) at 1 month ± 5 days.
Time Frame: at 1 month ± 5
Measure: Number; unit: participants
Arm/Group | Fondaparinux 1.5 mg/l
Number analyzed (Participants) | 442
participants | 3

5. Secondary Outcome: Death at 1 Month ± 5 Days
Description: Evaluate the total number of death at 1 month ± 5 days
Time Frame: 1 month ± 5 days
Measure: Number; unit: participants
Arm/Group | Fondaparinux 1.5 mg/l
Number analyzed (Participants) | 442
participants | 10

ADVERSE EVENTS:
Arm/Group | Fondaparinux 1.5 mg/l
Serious Adverse Events (participants affected / at risk) | 32/442
Other Adverse Events (participants affected / at risk) | 0/442
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fondaparinux 1.5 mg/l (N=442)
Hiatus hernia (Gastrointestinal disorders) | 1 (38)
Infarction mesenteric (Gastrointestinal disorders) | 1 (38)
Vomiting (Gastrointestinal disorders) | 1 (38)
gastrointestinal disorder NOS (Gastrointestinal disorders) | 1 (38)
Gastroduodenal hemorrhage (Gastrointestinal disorders) | 1 (38)
distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 (38)
proctorrhagia (Gastrointestinal disorders) | 1 (38)
Small intestine obstruction (Gastrointestinal disorders) | 1 (38)
Gastrointestinal obstruction NOS (Gastrointestinal disorders) | 1 (38)
Diarrhea, Clostridium difficile (Infections and infestations) | 1 (38)
septic shock (Infections and infestations) | 2 (38)
Bronchopulmonary infection (Infections and infestations) | 1 (38)
incision site infection (Infections and infestations) | 3 (38)
prosthesis fracture (Injury, poisoning and procedural complications) | 1 (38)
incision site hematoma (Injury, poisoning and procedural complications) | 3 (38)
anemia postoperative (Injury, poisoning and procedural complications) | 1 (38)
incision site inflammation (Injury, poisoning and procedural complications) | 1 (38)
femoral greater trochanter fracture (Injury, poisoning and procedural complications) | 1 (38)
Fracture of neck of femur (Injury, poisoning and procedural complications) | 1 (38)
deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 (38)
acute coronary syndrome (Cardiac disorders) | 2 (38)
acute myocardial infarction (Cardiac disorders) | 1 (38)
Atrial fibrillation paroxysmal (Cardiac disorders) | 1 (38)
cardio-respiratory failure (Cardiac disorders) | 1 (38)
transient cerebral ischemia (Nervous system disorders) | 1 (38)
ischemic strocke (Nervous system disorders) | 1 (38)
acute pulmonary edaema (Respiratory, thoracic and mediastinal disorders) | 2 (38)
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 (38)
Respiratort insufficiency (Reproductive system and breast disorders) | 1 (38)
mesenteric ischemia (Vascular disorders) | 1 (38)
malaise (General disorders) | 1 (38)
general physical health deterioration (General disorders) | 2 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No